CLINICAL TRIAL: NCT00624351
Title: A Phase IIb Randomized, Double-blind, Placebo-controlled, Dose and Dose Regimen-ranging Study of the Safety and Efficacy of Epratuzumab in Serologically-positive Systemic Lupus Erythematosus (SLE) Patients With Active Disease
Brief Title: Study of Epratuzumab in Serologically-positive Systemic Lupus Erythematosus (SLE) Patients With Active Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SL0007; 2007-002566-35 (EudraCT Number)
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Monoclonal antibody; B-Cell immunotherapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): Phosphate-buffered Saline (PBS) infusions at study weeks 0, 1, 2, and 3.
  Interventions: Other: Placebo
- EMAB 600mg (Experimental): 600 mg Epratuzumab infusions at study weeks 0, 1, 2, and 3.
  Interventions: Biological: Epratuzumab
- EMAB 100mg (Experimental): 100 mg Epratuzumab infusions at study weeks 0, and 2, and placebo at study weeks 1 and 3.
  Interventions: Biological: Epratuzumab; Other: Placebo
- EMAB 400mg (Experimental): 400 mg Epratuzumab infusions at study weeks 0, and 2, and placebo at study weeks 1 and 3.
  Interventions: Biological: Epratuzumab; Other: Placebo
- EMAB 1200mg (Experimental): 1200 mg Epratuzumab infusions at study weeks 0, and 2, and placebo at study weeks 1 and 3.
  Interventions: Biological: Epratuzumab; Other: Placebo
- EMAB 1800mg (Experimental): 1800 mg Epratuzumab infusions at study weeks 0, and 2, and placebo at study weeks 1 and 3.
  Interventions: Biological: Epratuzumab; Other: Placebo

INTERVENTIONS:
Biological: Epratuzumab — Epratuzumab at a concentration of 10 mg/mL prepared in 17.5 ml vials for slow intravenous infusion using only Phosphate buffered Saline (PBS) as a vehicle/buffer for the infusion procedure.
  Arms: EMAB 100mg; EMAB 1200mg; EMAB 1800mg; EMAB 400mg; EMAB 600mg
Other: Placebo — Phosphate-buffered Saline (PBS) infusion.
  Arms: EMAB 100mg; EMAB 1200mg; EMAB 1800mg; EMAB 400mg; Placebo

SUMMARY:
The primary objective of the study is to assess the dose response and the dose frequency of epratuzumab in patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

* Positive ANA result at visit 1
* Current diagnosis of systemic lupus erythematosus (SLE) by American College of Rheumatology revised criteria such that at least 4 of the 11 criteria are met
* Active moderate or severe SLE disease activity as demonstrated by British Isles Lupus Assessment Group (BILAG) A level disease activity in at least one body/organ system or BILAG B level disease activity in at least two body/organ systems if no BILAG A level disease is present
* If on antimalarials, dose regimen must be stable for 4 weeks prior to study entry.

Exclusion Criteria:

* Patients receiving any live vaccination within 2 weeks prior to visit 1 or during the course of the study
* Active severe SLE disease activity which involves the central nervous system (CNS) (defined by BILAG neurologic A level activity) including transverse myelitis, psychosis and seizures
* Active severe SLE disease activity which involves the Renal system (defined by BILAG renal level A activity or Grade III or higher World Health Organization (WHO) nephritis) or serum creatinine >2.5mg/dL or clinically significant serum creatinine increase within the prior 4 weeks or proteinuria >3.5gm/day
* Patients with a history of anti-phospholipid antibody syndrome AND use of oral anticoagulants or anti-platelet treatment
* Patients with a history of chronic infection, recent significant infection, or any current sign of symptom that may indicate an infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Response at Week 12 according to a combined response index | Week 12
  The combined response index incorporates the Bristish Isles Lupus Assessment Group (BILAG) assessment, the Systemic Lupus Eyrthematosus Disease Activity Index (SLEDAI), a physician's global assessment of disease activity, and treatment failure status.

SECONDARY OUTCOMES:
Response at Week 4 according to a combined response index | Week 4
  The combined response index incorporates the Bristish Isles Lupus Assessment Group (BILAG) assessment, the Systemic Lupus Eyrthematosus Disease Activity Index (SLEDAI), a physician's global assessment of disease activity, and treatment failure status.
Response at Week 8 according to a combined response index | Week 8
  The combined response index incorporates the Bristish Isles Lupus Assessment Group (BILAG) assessment, the Systemic Lupus Eyrthematosus Disease Activity Index (SLEDAI), a physician's global assessment of disease activity, and treatment failure status.
Response at Week 4 according to a combined response index involving Short Form-36 (SF-36) response | Week 4
  The combined response index incorporates the Bristish Isles Lupus Assessment Group (BILAG) assessment, the Systemic Lupus Eyrthematosus Disease Activity Index (SLEDAI), a physician's global assessment of disease activity, treatment failure status, and SF-36 response.
Response at Week 8 according to a combined response index involving Short Form-36 (SF-36) response | Week 8
  The combined response index incorporates the Bristish Isles Lupus Assessment Group (BILAG) assessment, the Systemic Lupus Eyrthematosus Disease Activity Index (SLEDAI), a physician's global assessment of disease activity, treatment failure status, and SF-36 response.
Response at Week 12 according to a combined response index involving Short Form-36 (SF-36) response | Week 12
  The combined response index incorporates the Bristish Isles Lupus Assessment Group (BILAG) assessment, the Systemic Lupus Eyrthematosus Disease Activity Index (SLEDAI), a physician's global assessment of disease activity, treatment failure status, and SF-36 response.
Improvement (yes/no) in British Isles Lupus Assessment Group (BILAG) at Week 4 | Baseline, Week 4
Improvement (yes/no) in British Isles Lupus Assessment Group (BILAG) at Week 8 | Baseline, Week 8
Improvement (yes/no) in British Isles Lupus Assessment Group (BILAG) at Week 12 | Baseline, Week 12
Improvement in British Isles Lupus Assessment Group (BILAG) at Week 24 | Baseline, Week 24
Change from baseline in total British Isles Lupus Assessment Group (BILAG) score at Week 12 | Baseline, Week 12
Change from baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) at Week 2 | Baseline, Week 2
Change from baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) at Week 4 | Baseline, Week 4
Change from baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) at Week 8 | Baseline, Week 8
Change from baseline in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) at Week 12 | Baseline, Week 12
Change from baseline in physician global assessment at Week 12 | Baseline, Week 12
Change from baseline in patient global assessment at Week 12 | Baseline, Week 12
Short Form-36 (SF-36) response at Week 2 | Baseline, Week 2
  SF-36 response is defined as no changes from baseline more negative than -0.8 in PCS or > -2.5 changes in any of the 8 domain scores.
Short Form-36 (SF-36) response at Week 4 | Baseline, Week 4
  SF-36 response is defined as no changes from baseline more negative than -0.8 in PCS or > -2.5 changes in any of the 8 domain scores
Short Form-36 (SF-36) response at Week 8 | Baseline, Week 8
  SF-36 response is defined as no changes from baseline more negative than -0.8 in PCS or > -2.5 changes in any of the 8 domain scores
Short Form-36 (SF-36) response at Week 12 | Baseline, Week 12
  SF-36 response is defined as no changes from baseline more negative than -0.8 in PCS or > -2.5 changes in any of the 8 domain scores
European Quality of Life-5 Dimensions (EQ-5D) score at Week 12 | Week 12
Time to first sustained British Isles Lupus Assessment Group (BILAG) response | From Baseline to Week 12
Time to enhanced British Isles Lupus Assessment Group (BILAG) response | From Baseline to Week 12
Treatment failure up to Week 12 | From Baseline to Week 12
  Treatment failure is defined as increase in (or addition of a new) immunosuppressive agent over baseline treatment levels, or any increase in corticosteroid baseline treatment level, or any IV, IA, or IM injections of corticosteroids.
Cumulative steroid dose at Week 12 | From Baseline to Week 12
Human anti-human antibodies (HAHA) levels at Week 12 | Week 12
Change from baseline in levels of circulating B cells at Week 12 | Baseline, Week 12
Change from baseline in levels of circulating T cells at Week 12 | Baseline, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (53):
- United States (19):
  - Birmingham, Alabama
  - Tucson, Arizona
  - La Jolla, California
  - Los Angeles, California
  - San Leandro, California
  - Denver, Colorado
  - Farmington, Connecticut
  - Aventura, Florida
  - Tampa, Florida
  - Baltimore, Maryland
  - Brooklyn, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Wilmington, North Carolina
  - Oklahoma City, Oklahoma
  - Dallas, Texas
  - Arlington, Virginia
  - Milwaukee, Wisconsin
- Belgium (2):
  - Brussels
  - Leuven
- Brazil (6):
  - Curitiba
  - Goiânia
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
  - Sorocaba
- Hong Kong (2):
  - Chai Wan
  - Shatin
- Hungary (2):
  - Debrecen
  - Zalaegerszeg
- India (6):
  - Bangalore
  - Hyderabad
  - Ludhiana
  - Madurai
  - Manipal
  - Nagpur
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Poland (5):
  - Elblag
  - Gmina Końskie
  - Lublin
  - Poznan
  - Torun
- Spain (3):
  - Barcelona
  - Santander
  - Valencia
- Ukraine (4):
  - Donetsk
  - Ivano-Frankivsk
  - Kiev
  - Lviv
- Birmingham, United Kingdom

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Wallace DJ, Kalunian K, Petri MA, Strand V, Houssiau FA, Pike M, Kilgallen B, Bongardt S, Barry A, Kelley L, Gordon C. Efficacy and safety of epratuzumab in patients with moderate/severe active systemic lupus erythematosus: results from EMBLEM, a phase IIb, randomised, double-blind, placebo-controlled, multicentre study. Ann Rheum Dis. 2014 Jan;73(1):183-90. doi: 10.1136/annrheumdis-2012-202760. Epub 2013 Jan 12. PMID 23313811